CLINICAL TRIAL: NCT06240702
Title: The Effect of Early Cardiopulmonary Telerehabilitation on Exercise Capacity, Cardiac Function, Quality of Life and Emotional Status in Coronary Bypass Surgery Patients
Brief Title: Effects of Early Telerehabilitation in Coronary Artery Bypass Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Muammer Corum, Lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-SSHMYO-FP-MC-01
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease; Cardiac Disease
Keywords: Coronary Artery Bypass; Cardiac Rehabilitation; Sleep Hygiene; Telerehabilitation; Exercise
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Sleep Hygiene; Motor Activity

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled clinical trial with 2 groups, experimental and control. The experimental group will be treated with telerehabilitation while the control group will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation Group (Experimental): Patients in the experimental group will be included in the face-to-face Phase I rehabilitation program until discharge and in the Phase II telerehabilitation program and sleep hygiene training for 3 weeks after discharge. Respiratory exercises will be performed as part of the phase I rehabilitation program until the patients are discharged. In addition, active range of motion and mobility exercises in bed, sitting position and standing, increasing distance walking and stair ascent and descent training will be provided. During the sessions, the patient's vital signs and clinical status will be monitored with a finger pulse oximeter and a blood pressure measuring device according to the patient's perceived degree of difficulty (Borg Scale). As part of the Phase II telerehabilitation program, respiratory exercises, calisthenic exercises and gait training will be performed.
  Interventions: Other: Telerehabilitation Group
- Control Group (No Intervention): Patients in the control group will be included in the face-to-face Phase I rehabilitation program until discharge and no intervention will be made after discharge. Until the patients in the control group are discharged, respiratory exercises will be performed as in the experimental group within the scope of the phase I rehabilitation program. In addition, active range of motion and mobility exercises in bed, sitting position and standing, increasing distance walking and stair ascent and descent training will be provided. During the sessions, the patient's vital signs and clinical status will be monitored with a finger pulse oximeter and a blood pressure measuring device according to the patient's perceived degree of difficulty (Borg Scale).

INTERVENTIONS:
Other: Telerehabilitation Group — Unlike the control group, the experimental group will be given a phase II telerehabilitation program and sleep hygiene training for 3 weeks after discharge. Within the scope of the Phase II telerehabilitation program, breathing exercises and calisthenic exercises will be performed at increasing intensity according to the patient's tolerance, 3 days a week for 3 weeks. In addition, walking training will be continued over increasing distances. In addition, it will be aimed to increase sleep quality by giving a sleep hygiene education brochure to the patients in the experimental group. During the sessions, the vital signs and clinical status of the patients will be monitored according to the severity level determined by the finger pulse oximeter device, digital blood pressure monitor, perceived difficulty level (Borg Scale) and maximum heart rate. In addition, patients will be kept in a diary to monitor their compliance with the treatment program.
  Arms: Telerehabilitation Group

SUMMARY:
The aim of this study was to investigate the effects of phase I and early phase II rehabilitation with telerehabilitation method and sleep hygiene training on physical capacity, cardiac functions, anxiety level, quality of life and sleep quality in patients undergoing coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
Coronary artery disease is one of the most important diseases affecting quality of life in recent years. Coronary artery bypass graft surgery (CABGC), one of the methods used in the treatment of this disease, is widely accepted as a common operation. However, both the surgical intervention and the cardiac and pulmonary complications caused by coronary artery disease, such as decreased physical capacity, decreased quality of life and sleep quality, and restriction in functional activities make it difficult to return to pre-disease level. Today, it is a scientific fact that cardiac and pulmonary rehabilitation applied at the earliest period following surgical treatment reduces the risk of mortality and morbidity, prevents complications and facilitates return to daily life. In fact, it is now a necessity to evaluate and treat patients comprehensively in many aspects such as nutrition, sleep quality and psychological status with a holistic approach. Today, applications that bring together healthcare personnel and patients in a virtual environment such as telemedicine, telerehabilitation and mobile-health, which have been widely used in different medical and health fields, especially after the coronavirus-19 pandemic, have gained importance. Telerehabilitation has advantages in different fields such as neurological, orthopedic, cardiac and pulmonary rehabilitation, such as the ability of the physiotherapist to follow the patient remotely, to apply the rehabilitation program, and to be accessible at any time. In addition, it is stated in the literature that it has mitigating effects on the patient's dependency and health costs, such as eliminating the need for the patient to travel to the center and reducing the need for caregivers. When the literature is examined, it is seen that there are few cardiac and pulmonary rehabilitation applied with telerehabilitation method in the postoperative period in coronary artery bypass graft surgery patients. In addition, there is no study in the literature examining the effect of sleep hygiene training in addition to telerehabilitation on these patients. Therefore, this study aimed to contribute to the literature as an original study by examining the effects of cardiopulmonary rehabilitation and sleep hygiene training applied for 4 weeks with the telerehabilitation method, which is a current approach, on patients who underwent coronary artery bypass graft surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are class 2-3 according to the New York Heart Association (NYHA)
* Participants had an ejection fraction >40%
* If the participant has had a myocardial infarction (MI), 7 days have passed since the MI
* Low-medium risk group patients as a result of Euroscore evaluation (0-2 low risk, 3-5 medium risk, 6< high)
* Patients with adequate cognition-perception level (Mini mental test score of 24 and above)
* Individuals who are not diagnosed with sleep disorders for any reason
* Having the knowledge to make video calls with a smart phone
* Declaring that you wish to participate in the study with written consent

Exclusion Criteria:

* Aneurysm history
* Patients with advanced left ventricular dyskinesia
* Patients with neurological orthopedic comorbid diseases
* Presence of any defect in the rib cage
* Patients with Chronic Obstructive Pulmonary Disease (COPD)
* Patients hospitalized for a long time (6 months and more)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
6 minute walk test (6MWT) | four weeks
  The test is performed in a closed area, on a flat surface 30 meters long (every 3 meters is marked), under the supervision of a physiotherapist. Dyspnea and fatigue of the patients are questioned during the 6MWT and the values before and after the test are recorded. At the end of 6 minutes, the total distance walked by the patient is recorded in meters. Studies have shown that a 6-minute walking distance of less than 350 meters is a predictor of mortality in cardiopulmonary diseases.
Duke Activity Status Scale | four weeks
  This 12-question index helps to calculate the metabolic equivalent of task (MET) used in daily life. 1 MET represents the resting Oxygen consumption of a 40-year-old 70 kg person at rest, which is normally 3.5 ml/kg/min. According to this index; self-care, eating, dressing, going to the toilet, short walks inside the house, short walks outside, light housework, between 1-4 METs; climbing hills or stairs, fast walking, short jogging, heavier work at home, light sports, between 4-10 METs; Heavy sports such as swimming, tennis are evaluated above 10 METs. The approximate values obtained according to the answers to the questions asked are classified as follows; Excellent if >7 MET 4-7 MET is Moderate <4 MET indicates a poor or uncertain prognosis.
State Trait Anxiety Inventory | four weeks
  The Turkish version of the State Trait Anxiety Inventory (STAI) will be used to assess the anxiety level of the subjects. The STAI consists of 2 parts, the state anxiety scale and the trait anxiety scale, and a total of 40 questions. When answering the state anxiety scale, patients are asked to select one of the options 'not at all', 'a little', 'a lot' and 'completely' according to the severity of the feelings, thoughts and behaviors expressed by the items; when answering the trait anxiety scale, patients are asked to mark one of the options 'almost never', 'sometimes', 'most of the time' and 'almost always' according to the frequency of the feelings, thoughts and behaviors expressed by the items. High scores indicate a high level of anxiety. Turkish validity and reliability studies have been conducted.
Pittsburgh Sleep Quality Index (PSQI) | four weeks
  PSQI was adapted into Turkish by Agargun et al. (1996). PSQI evaluates sleep quality in the last month. 19 of the total 24 questions included in PSQI are self-report questions. 5 questions are answered by the spouse or a roommate. The last 5 questions mentioned are used only for clinical information and are not included in the scoring. The 18 items included in the scoring are grouped into 7 component scores. Some of the components are specified with a single item, while others are obtained by grouping several items. Each item is evaluated on a scale of 0-3 points. The sum of the 7 component scores gives the total PSQI score. The total score has a value between 0-21. A high total score indicates poor sleep quality.

SECONDARY OUTCOMES:
Echocardiography | four weeks
  The term echocardiography covers all imaging techniques in which the heart is examined with ultrasound, such as pulsed and continuous wave Doppler, color Doppler and tissue Doppler imaging (TDI: tissue doppler imaging). Echocardiography is an easily accessible, non-invasive, rapid and safe method that provides comprehensive information on cardiac anatomy (volumes, geometry, mass), wall motion and valve function.
Left Ventricular Dysfunction Scale (LVD-36) | four weeks
  The Left Ventricular Dysfunction (LVD-36) Scale was developed by O'Leary and Jones (2000) to measure the effect of left ventricular dysfunction on daily life and well-being in patients with heart failure. This scale; It consists of a total of 36 statements asked to determine the problems caused by heart disease. Statements are presented to patients with two options: true or false. The correct answers given are added up and the total number of correct answers is expressed as a percentage. Scores from the scale are between "0-100", with "100 points" taken from the scale being considered the worst score and "0 points" being considered the best score. As the score of the scale increases, the quality of life decreases. The Turkish validity and reliability study of the LVD-36 scale was conducted by Özer and Argon (2005).
Minnesota Living With Heart Failure Questionnaire | four weeks
  It is a quality of life survey consisting of 21 questions and two dimensions (physical and emotional sub-dimensions) specific to Heart Failure patients. It was designed by Thomas Rector in 1984 to measure the impact of heart failure and its treatment on an individual's quality of life. The survey was prepared in Likert type. The survey assesses the impact of common physical symptoms such as shortness of breath, fatigue, peripheral edema, symptoms of anxiety and depression. In addition, it aims to measure the effects of physical and social functioning in heart failure. The lowest score that can be obtained from the scale is 5 and the highest score is 105. The Turkish adaptation was made by Uzunhasanoglu in 2013.
Modified Medical Research Council Dyspnea Scale | four weeks
  The scale used to evaluate patients' shortness of breath classifies it from stage 1 to stage 5 to determine the severity of shortness of breath.
Hand Grip Strength Assessment | four weeks
  Upper extremity muscle strength will be evaluated with a hand dynamometer. It has been reported that hand grip strength is not only correlated with upper extremity muscle strength, but also with general body muscle strength and pulmonary muscle strength. Test; It will be made in the sitting position, which is the standard position recommended by the American Association of Hand Therapists, with the shoulder in adduction and neutral rotation, the elbow in 90° flexion, the forearm in middle rotation, and the wrist in neutral. Three measurements will be made, the average will be taken and recorded as kg/F. In addition, pinch grip strength will be measured in the same way with a pinch meter type dynamometer.
30-second sit-to-stand test | four weeks
  This test reflects the strength of the lower extremities. The individual sits on the middle part of the chair, which has no armrests and a sitting height of 43.18 cm, with his back upright and straight, his arms crossed in front, and his feet flat on the floor. It stands up and sits down fully upon the start command. Count the number of times he stands up fully in 30 seconds.
Body Weight | four weeks
  Participants' body weight will be recorded as demographic data in kg unit.
Body height | four weeks
  The height of the participants will be recorded as demographic data in meters unit.
Body Mass Index | four weeks
  Participants' body mass index will be recorded as demographic data in kg/m² unit.
Heart Rate | four weeks
  Participants' heart rates before and after the intervention will be recorded in beats/minute.
Blood Pressure | four weeks
  The blood pressure of the participants before and after the intervention will be recorded in mmHg.
Respiratory Frequency | four weeks
  The respiratory frequency of the participants before and after the intervention will be recorded as breaths/minute.
Oxygen Saturation | four weeks
  The oxygen saturation of the participants before and after the intervention will be recorded as SaO₂(%).

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Dogan, Assoc. Prof., Study Director — Necmettin Erbakan University Faculty Member
Locations (1):
- Necmettin Erbakan University Faculty of Medicine, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No